CLINICAL TRIAL: NCT04639869
Title: Open-label, Randomized, Single Dose, 4period, Replicated, Cross-over Trial to Assess the Bioequivalence of Feniramidol HCl 400 mg Film Tablet in Comparison With Cabral 400 mg Film Tablet in Healthy Male Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Feniramidol HCl 400 mg Film Tablet (Pharmactive, Turkey) Under Fed Conditions
Acronym: PHENYRAMIDOL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Collaborators: Novagenix Bioanalytical Drug R&D Center (Network); Farmagen Ar-Ge Biyot. Ltd. Sti (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NOV2019/01864
Record Dates: First submitted 2020-09-29; First posted 2020-11-23 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2020-11

CONDITIONS: Bioequivalence
Keywords: Phenyramidol; Pharmactive Ilaç San.ve Tic. A.S
MeSH Terms: interventions — Motion Pictures

STUDY DESIGN:
Intervention Model Description: Full replicate cross-over bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phenyramydol then Cabral (Experimental): Participants first receive Phenyramydol HCl 400 mg Film Tablet manufactured by Pharmactive Ilac San ve Tİc A.S. in fed state. After a wash out period of 7 days, they then received Cabral 400 mg Film Tablet manufactured by Recordati Ilac San ve Tİc A.S. in fed state
  Interventions: Drug: Phenyramydol HCl 400 mg Film Tablet; Drug: Cabral 400 mg Film Tablet
- Cabral then Phenyramydol (Active Comparator): Participants first receive Cabral 400 mg Film Tablet manufactured by Recordati Ilac San ve Tİc A.S. in fed state. After a wash out period of 7 days, they then received Phenyramydol HCl 400 mg Film Tablet manufactured by Pharmactive Ilac San ve Tİc A.S.in fed state
  Interventions: Drug: Phenyramydol HCl 400 mg Film Tablet; Drug: Cabral 400 mg Film Tablet
- Phenyramydol then Cabral Replicate (Experimental): Participants first receive Phenyramydol HCl 400 mg Film Tablet manufactured by Pharmactive Ilac San ve Tİc A.S. in fed state. After a wash out period of 7 days, they then received Cabral 400 mg Film Tablet manufactured by Recordati Ilac San ve Tİc A.S. in fed state
  Interventions: Drug: Phenyramydol HCl 400 mg Film Tablet; Drug: Cabral 400 mg Film Tablet
- Cabral then Phenyramydol Replicate (Active Comparator): Participants first receive Cabral 400 mg Film Tablet manufactured by Recordati Ilac San ve Tİc A.S. in fed state. After a wash out period of 7 days, they then received Phenyramydol HCl 400 mg Film Tablet manufactured by Pharmactive Ilac San ve Tİc A.S.in fed state
  Interventions: Drug: Phenyramydol HCl 400 mg Film Tablet; Drug: Cabral 400 mg Film Tablet

INTERVENTIONS:
Drug: Phenyramydol HCl 400 mg Film Tablet — Phenyramydol HCL 400 mg Film Tablet contains 400 mg phenyramydol manufactured by Pharmactive Ilac.San ve Tic A.S
  Other Names: Test Phenyramydol
Drug: Cabral 400 mg Film Tablet — Cabral 400 mg Film Tablet 400 mg phenyramydol manufactured by Recordati Ilac SAn ve Tic A.S.
  Other Names: Reference Phenyramydol

SUMMARY:
OPEN-LABEL, RANDOMISED, SINGLE ORAL DOSE, FOUR-PERIOD, REPLICATED, CROSS-OVER TRIAL TO ASSESS THE BIOEQUIVALENCE OF FENIRAMIDOL HCl 400 MG FILM TABLET (TEST DRUG) IN COMPARISON WITH CABRAL 400 MG FILM TABLET (REFERENCE DRUG) IN HEALTHY MALE SUBJECTS UNDER FED CONDITIONS

DETAILED DESCRIPTION:
Phenyramidol shows its muscle relaxant activity by interneuronal blockage without disrupting neuromuscular function. Thus, it relieves muscle spasm, and breaks pain-spasm chain by blocking polisynaptic reflexes in the brain and medulla spinalis. It does not affect monosynaptic reflexes.

Phenyramidol has a very high analgesic effect than aspirin and close to codeine. It used in the treatment of acute and chronic human musculoskeletal system pains as muscle relaxant and analgesic.

Pharmacokinetics Phenyramidol reaches maximum plasma concentration in an hour (0.25-1) after absorption from gastrointestinal tract. It is widely distributed in skeletal muscles and involved in circulatory system very slowly.

Studies have shown that cytochrome P450 enzymes are effective in phenyramidol metabolism. It is conjugated with glucuronic acid in the liver and it is excreted as glucuronide conjugates from the urinary tract. The drug is eliminated from the bile and the bacterial glucuronidase enzymes make the glucuronide conjugate of phenyramidol free. The drug enters enterohepatic circulation and is excreted by faeces. Its elimination half-life is 1-2 hours.

Indications Phenyramidol is indicated in the symptomatic treatment of acute painful muscle spasms associated with musculoskeletal system.

ELIGIBILITY:
Inclusion Criteria:

Only volunteers fulfilling all of the following criteria should be enrolled in the present trial:

1. Healthy Caucasian male subjects aged between 18 and 55 years,
2. Non smokers or smoking maximum 5 cigarettes a day, those who won't smoke or drink coffee during each study period,
3. Negative alcohol breath test results,
4. Normal physical examination at screening visit,
5. Having the Body Mass Index ranged between 18.5-30 kg/m2 (see Appendix I) which is in the desirable range according to the age,
6. Ability to communicate adequately with the investigator himself or his/her representatives,
7. Ability and agreement to comply with the study requirements,
8. Normal blood pressure and heart rate measured under stabilised conditions at the screening visit after at least 5 minutes of rest under supine position: SBP within 100 to 140 mmHg, DBP within 60 to 90 mmHg and HR within 50 to 90 bpm,
9. Normal/ acceptable 12-lead electrocardiographic results at least after 5 minutes of rest,
10. Laboratory results within normal range or clinically non-significant (CBC, glucose, urea, uric acid, creatinine, estimated GFR (eGFR), total bilirubin, sodium, potassium, calcium, chloride, SGOT (AST), SGPT (ALT), GGT, alkaline phosphatase, total protein and urinalysis), drug addiction scanning in urine results in negative (amphetamine, barbiturate, benzodiazepine, cannabinoid, cocaine, opiate),
11. Understanding of the study and agreement to give a written informed consent according to section 20.3.

Exclusion Criteria:

Volunteers presenting any of the following exclusion criteria will not be included in the trial:

1. Who have atopic constitution or asthma and/or known allergy for phenyramidol HCl or any other ingredients of the products.
2. Any history or presence of clinical relevance of cardiovascular, neurological, musculoskeletal, haematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolism or psychiatric disease, any type of porphyria.
3. Symptomatic or asymptomatic orthostatic hypotension at screening or before the first drug administration defined by a decrease of SBP more than 20 mmHg or DBD more than 10 mmHg occurs between sitting/supine to standing position subject will be excluded (if it deemed necessary by the investigator).
4. Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or except herniotomy.
5. Subjects who have given more than 400 mL blood within the last two months before the first drug administration and subjects who have participated to any drug research within the last two months before the first drug administration.
6. Subjects suspected to have a high probability of non-compliance to the study procedure and/or completion of the study according to the investigator's judgement.
7. Subjects who used any of prescribed systemic or topical medication (including OTC medication) within 2 weeks (or six elimination half lives of this medication, whichever is longer) before the initiation of the study (except single doses of analgesics which have no drug interaction with study product).
8. Use of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
9. History of allergic response to heparin.
10. Subjects who have any chronic disease which might interfere with absorption, distribution, metabolism or excretion of the drug.
11. Subjects who regular consumed of beverages or food containing methylxanthines (e.g. coffee, tea, cola, caffeine, chocolate, sodas,) equivalent to more than 500 mg methylxanthines per day.
12. Subjects who has taken any grapefruit or grapefruit juice during 7 days prior to drug administration, during the study, or during the washout periods.
13. History of drug abuse.
14. History of alcohol abuse and/or regular use of more than 2 units of alcohol per day or 10 units per week and/or positive alcohol breath test results (Note: one unit of alcohol equals 250 mL beer, 125 mL wine or 25 mL spirits).
15. Positive blood test for HBV, HCV and HIV.
16. Who have relationship to the investigator.
17. Who are not suitable to any of inclusion criteria.
18. History of difficulty of swallowing.
19. Intake of depot injectable solutions (including study medications) within 6 months before start of the study.
20. Intake of enzyme-inducing, organotoxic or long half-life drugs within 4 weeks before start of the study.
21. Special diet due to any reason, e.g. vegetarian.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 to 10 hours post-dose
  Cmax of phenyramydol will be obtained from plasma concentrations
AUCt-last | 0 to 10 hours post-dose
  AUC0-tlast of phenyramydol will be obtained from plasma concentrations
AUC0-inf | 0 to 10 hours post-dose
  AUC0-inf of phenyramydol will be obtained from plasma concentrations

SECONDARY OUTCOMES:
tmax | 0 to 10 hours post-dose
  tmax of phenyramydol will be obtained from plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Muradiye Nacak, MD,PhD, Principal Investigator — Farmagen Ar-Ge Biyot. Ltd. Sti; Taner Ezgi, MD, Study Chair — Farmagen Ar-Ge Biyot. Ltd. Sti; Hakan Gürpınar, MSc, Study Director — Pharmactive İlaç San.ve Tic.A.S
Locations (1):
- Novagenix Drug R&D Center, Akyurt, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04639869/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04639869/ICF_001.pdf